CLINICAL TRIAL: NCT03199742
Title: Evaluation of a Mobile Phone App for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Owen, Clinical Psychologist, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-31533
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Stress Disorders, Post-Traumatic; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive one of 2 forms of the mobile phone application being tested in this study: with and without personalized coaching. Among those who receive coaching, participants will receive either peer-based coaching messages, clinician-based coaching messages, or automated messages.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PTSD Coach with no Coaching (Active Comparator): Participants will receive the PTSD coach mobile app.
  Interventions: Behavioral: Active Comparator
- PTSD Coach with Peer Coaching (Experimental): Participants will receive the PTSD Coach + mobile app which will provide routine, personalized coaching for 8 weeks from a Veteran peer.
  Interventions: Behavioral: Personalized App Coaching
- PTSD Coach with Clinician coaching (Experimental): Participants will receive the PTSD Coach + mobile app which will provide routine, personalized coaching for 8 weeks from a clinical psychologist.
  Interventions: Behavioral: Personalized App Coaching
- PTSD Coach with Automated Coaching (Experimental): Participants will receive the PTSD Coach + mobile app which will provide automated, personalized coaching for 8 weeks.
  Interventions: Behavioral: Personalized App Coaching

INTERVENTIONS:
Behavioral: Personalized App Coaching — All coaching messages will be based on how each participant responds to baseline survey questionnaires and how they interact with the experimental mobile phone application during the course of the study. Participants will be provided with feedback about recent progress & use of the app, information about coping strategies provided by the app, and a recommendation for making the best use of the app over the subsequent few days.
  Arms: PTSD Coach with Automated Coaching; PTSD Coach with Clinician coaching; PTSD Coach with Peer Coaching
Behavioral: Active Comparator — Mobile phone application providing extensive information about PTSD and treatment, tools for managing PTSD symptoms, self-monitoring using the PTSD Checklist, and resources for obtaining support.
  Arms: PTSD Coach with no Coaching

SUMMARY:
The purpose of this study is to evaluate a mobile phone app designed to help Veterans with PTSD. Participants in this study will be randomized to receive one of 2 possible mobile phone apps. The term "randomized" means that which app a participant receives will not be based on any characteristic or behavior of the participant, but will be determined solely by chance like a flip of a coin.

DETAILED DESCRIPTION:
Participants will receive access to the mobile app "PTSD Coach". Participants will be randomized (by computerized coin flip) to one of two versions of the mobile app. All versions of the app will provide comprehensive information and tools for managing trauma symptoms, but one version of the app will provide personalized, confidential coaching messages delivered by either a Veteran peer or clinical psychologist. Participants will be asked to complete an online survey before using the mobile phone application and again 8 weeks later. Participants will be provided with the option to complete a telephone interview after 8 weeks of using the mobile phone application. To be eligible, participants must be a U.S. military Veteran, age 18 or older, have received a previous diagnosis of PTSD, and own an iPhone or iPad device.

ELIGIBILITY:
Inclusion Criteria:

* U.S. military Veteran
* age 18 or older
* previously diagnosed with PTSD
* own an iPhone or iPad device

Exclusion Criteria:

* no previous history of PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist 5 | 8 weeks
  Measures symptoms of post-traumatic stress disorder
Functional Well-Being | 8 weeks
  Measures functional well-being of Veterans across a number of domains, including self-care, romantic relationships, work, family functioning, and parenting. Subscale scores will be aggregated to create a summary score for this measure.
Engagement with the Application | 8 weeks
  Objectively-measured engagement with the intervention (# sessions)

SECONDARY OUTCOMES:
Self-Efficacy for Coping | 8 weeks
  Self-efficacy for managing symptoms of PTSD using an author-constructed outcome measure.
Perceived Helpfulness of Intervention | 8 weeks
  How helpful the intervention was for providing information and tools for managing PTSD.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System Menlo Park Division, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No